CLINICAL TRIAL: NCT00537355
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of TOLAMBA™ in the Control of Symptoms of Ragweed-Allergic Rhinitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: An Evaluation of the Efficacy and Safety of TOLAMBA™ for Ragweed-Allergic Rhinitis in an Environmental Exposure Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DV1-SAR-11
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: ragweed; ragweed allergy; allergy; allergies; allergic; seasonal allergic rhinitis; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Rhinitis, Allergic | interventions — Histamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOLAMBA™ (Active Comparator)
  Interventions: Biological: Amb a 1 Immunostimulatory Oligoribonucleotide Conjugate
- Histamine (Sham Comparator): Histamine simulates mild redness/swelling effect seen with active comparator, TOLAMBA™. Prevents study staff from easily identifying subjects who received active comparator.
  Interventions: Drug: Histamine

INTERVENTIONS:
Biological: Amb a 1 Immunostimulatory Oligoribonucleotide Conjugate — 6 weekly subcutaneous injections (escalating doses of 3 mcg to 30 mcg)
  Other Names: TOLAMBA™
  Arms: TOLAMBA™
Drug: Histamine — 6 weekly subcutaneous injections (escalating doses of 0.22 mcg to 1.1 mcg)
  Other Names: Histatrol
  Arms: Histamine

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, parallel-group, multicenter study. After passing the initial Screening Visit, subjects will be in the environmental exposure chamber(EEC), a room with a controlled amount of ragweed pollen, for 4 hours each day on 4 consecutive days. At the last visit, subjects who have achieved a minimum Total Nasal Symptom Score (TNSS) will be randomized to receive either TOLAMBA or placebo treatments. Subjects will receive 6 weekly subcutaneous (under the skin) injections of the study drug. About three weeks after the last injection, subjects will be asked to be in the EEC for 2 consecutive days (Visits 11 and 12, Days 60 and 61). Approximately 3 weeks after Visit 12 (Day 61), the subjects will again be in the EEC for 4 consecutive days (Visits 13-16, Days 82-85).

During all EEC visits, the subjects will be exposed to ragweed pollen at an average concentration of 3500 ± 500 pollen grains per cubic meter. Each EEC visit will last 4 hours. During each EEC visit, patients will be asked to record symptom scores for nasal and non-nasal symptoms at scheduled time points.

The total duration of a subject's participation in this study is expected to be a minimum of 85 days.

DETAILED DESCRIPTION:
Ragweed allergy is the most common seasonal allergy in North America. Allergen immunotherapy is a therapeutic option for patients who have allergy symptoms that cannot be adequately controlled by avoidance of the allergen or medication. It may also be appropriate for those who cannot tolerate their medications due to side effects or have difficulties with medication compliance.

This will be a randomized, double-blind, placebo-controlled, parallel-group, multicenter study. After passing the initial Screening Visit, subjects will be in the environmental exposure chamber(EEC), a room with a controlled amount of ragweed pollen, for 4 hours each day on 4 consecutive days. At the last visit, subjects who have achieved a minimum Total Nasal Symptom Score (TNSS) will be randomized to receive either TOLAMBA or placebo treatments. Subjects will receive 6 weekly subcutaneous (under the skin) injections of the study drug. About three weeks after the last injection, subjects will be asked to be in the EEC for 2 consecutive days (Visits 11 and 12, Days 60 and 61). Approximately 3 weeks after Visit 12 (Day 61), the subjects will again be in the EEC for 4 consecutive days (Visits 13-16, Days 82-85).

During all EEC visits, the subjects will be exposed to ragweed pollen at an average concentration of 3500 ± 500 pollen grains per cubic meter. Each EEC visit will last 4 hours. During each EEC visit, patients will be asked to record symptom scores for nasal and non-nasal symptoms at scheduled time points.

The total duration of a subject's participation in this study is expected to be a minimum of 85 days.

Comparison: Allergy symptoms of subjects treated with TOLAMBA™ compared with subjects treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to give signed informed consent, and must have provided this consent.
* Has a clinical history of seasonal allergic rhinitis with seasonal nasal allergy symptoms during each of the last 2 ragweed allergy seasons.
* Has documentation of a positive skin test to ragweed allergen within 12 months of screening.
* Has minimum qualifying symptom scores at the last visit of the Pre-Treatment EEC sessions (Visit 5, Day 4).
* If female of childbearing potential, is not pregnant and is consistently using an acceptable birth control method.
* Is normally active and otherwise judged to be in good health on the basis of medical history, physical examination and routine laboratory tests.

Exclusion Criteria:

* A woman who is pregnant, breastfeeding, or planning a pregnancy.
* Has a history of more than mild asthma that requires the use of a daily inhaled or oral corticosteroid, leukotriene inhibitor, or cromolyn; or a daily inhaled short or long acting β-agonist.
* Has had any hospital admissions for asthma, a recent (within the past 12 months)asthma exacerbation that required either oral or inhaled corticosteroids, or a prior history of unstable asthma.
* Has received immunotherapy within the last 2 years that has contained ragweed pollen extract.
* Has previously participated in a clinical trial with TOLAMBA or another ragweed-based immunotherapy.
* Has received immunotherapy for any allergens within 30 days prior to Visit 1.
* Has the need for use of antihistamines or corticosteroids on a regular basis (systemic or topical).
* Has received anti-immunoglobulin E (IgE) antibody (Xolair®) within the past 12 months.
* Is currently taking monoamine oxidase (MAO) inhibitors.
* Has taken any systemic corticosteroids, immunomodulators, or immune suppressive medications within 4 weeks prior to Visit 1.
* Has taken any antihistamine within 7 days prior to Visit 1 skin testing.
* Requires use of β-adrenergic blockers or other agents that may interfere with the use of adrenaline.
* Known current alcohol or drug abuse.
* Current participation in another clinical study involving an investigational drug or device, or participation in such a study within 30 days prior to Visit 1.
* Has a history of generalized anaphylaxis requiring medical attention.
* Has moderate or severe allergy symptoms at Visit 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 3 months

SECONDARY OUTCOMES:
Total Non-Nasal Symptom Score (TNNSS) | 3 months
Total Symptom Score (TSS) | 3 months
quality of life questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, DPhil, Study Director — Dynavax Technologies Corporation
Locations (6):
- Canada (6):
  - Allied Research International Inc., Mississauga, Ontario
  - Alpha Medical Research Inc., Mississauga, Ontario
  - Allergy & Asthma Research Centre, Ottawa, Ontario
  - Division of Clinical Immunology and Allergy, The McGill University Health Centre, Montreal, Quebec
  - Anapharm, Montreal, Quebec
  - Centre De Recherche Appliquée en Allergie De Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
The IND for Tolamba was withdrawn. There is no intention to conduct clinical studies with this compound. All studies were conducted in Canada, no U.S. sites participated in study. CT PRS states "DR" status will be removed from study. 3/1/2017 - no update

REFERENCES:
- [Derived] Campbell JD, Buchmann P, Kesting S, Cunningham CR, Coffman RL, Hessel EM. Allergen-specific T cell responses to immunotherapy monitored by CD154 and intracellular cytokine expression. Clin Exp Allergy. 2010 Jul;40(7):1025-35. doi: 10.1111/j.1365-2222.2010.03505.x. Epub 2010 Apr 13. PMID 20412135
- See also: sponsor website — http://www.dynavax.com